CLINICAL TRIAL: NCT04809194
Title: Digital Signals of Stress in Crohn's: Forecasting Symptom Transitions
Brief Title: Stress in Crohn's Disease
Status: Completed | Type: Observational
Sponsor: 4YouandMe (Other)
Collaborators: Evidation Health (Industry); Vector Institute of Artificial Intelligence (Unknown); Icahn School of Medicine at Mount Sinai (Other); Oxford University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 4UCROHNS01
Record Dates: First submitted 2021-03-19; First posted 2021-03-22 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Crohn Disease
Keywords: Digital health, Crohn's disease, Wearable technology
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stool sample to measure calprotectin using IBDoc Kits
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
There is little information on how Crohn's disease progresses in between a patient's clinic visits and how stress impacts symptom change including flare-ups. The purpose of this research study is to see if digital tools like smartphones, and wearable devices are helpful in finding out new information that may explain fluctuation in symptoms. This study is a feasibility study that will try to identify biomarkers, collected through a smartphone app and wearable devices paired with clinical information collected during clinic visits to track participants' overall health for 6 to 12 months. The data collected will be used to identify and predict symptoms associated with Crohn's disease flare ups. The aim of this work is to inform knowledge of what triggers Crohn's disease worsening that might lead to advances in management.

DETAILED DESCRIPTION:
Crohn's disease is a relapsing and remitting condition, and each patient's course through their illness is unique across a range of life events. In people with Crohn's disease as with the general population, there are relationships between external stressors, internal emotional states and psychological experiences, such as how one experiences illness. The output of these aforementioned states has very rarely been studied in multiple body-systems, particularly in diseases of the gut which has many connections to the nervous system and uses many of the same chemical signalling pathways in the brain.

Through close and continuous measurement of physiological, behavioral, and experiential information we will track participants over time by using smartwatches, smart rings, and smartphones on a cohort of over 200 patients with Crohn's disease in the United States and the United Kingdom to build a longitudinal model of each participant's disease. We will measure the patient's stress response using these tools to generate manual and passive data. The first is a customized application installed on the participant's own phone, which will track both passive sensor measurement and participant-generated active-task data. Additionally, a "smart" wristwatch and "smart" finger-ring wearable devices will be given to the participant for the duration of the study. The multimodal acquisition of periodic subjective data and continuous objective data collected by the two wearable devices will constitute an unprecedented comprehensive picture of each individual, their disease trajectory, and its connection to their stress response. All these signals will be anchored to clinic visits. As a result of following several hundred participants over the course of six to nine months, meaningful models of each individual's unique disease course as well as generalizable models that classify individuals into definable similar trajectories will be developed. This study will explore the feasibility and provide the direction for the studies needed to build out comprehensive individual forecasting tools for people with Crohn's disease to manage their own conditions.

Ultimately, providing this early warning information from wearables directly to the individual will enable each patient to adapt aspects of their lifestyle, including exposure to modifiable stress, to prevent negative clinical changes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Crohn's disease previously established by endoscopy, imaging, and/or histology
* Disease of the small bowel, large bowel, or both large and small bowel
* Needs to have at least one flare in the last 12 months while on current therapy
* Subjects may be on no treatment or may have concurrent treatment with 5-aminosalicylates, antibiotics, corticosteroids, thiopurines, methotrexate or biologic therapies, including infliximab, adalimumab, certolizumab pegol, vedolizumab, or ustekinumab
* Disease level, see stratified enrollment below
* Subjects must have a personal cell phone that is an iPhone SE or newer and be willing to upgrade to the most recent iOS operating system and use their phone for study. This includes a willingness to download and use the study applications and sync their phone with the necessary study devices.

Exclusion Criteria:

* Imminent indication for surgery, such as small bowel obstruction or abscess, or surgery in the past 4 weeks
* More than 100 cm of small bowel resected
* Dependence on chronic enteral supplementation or parenteral nutrition or fluids
* Ileostomy or Colostomy (some of the outcome measures do not apply as cannot count # bowel movements)
* History of asymptomatic Crohn's disease for the last 2 years
* Current use of investigational therapy
* Self-reported pregnancy or intent to become pregnant during the study period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Crohn's disease attending clinics from the Icahn School of Medicine at Mount Sinai (n=140) and the Oxford Nuffield Department of Medicine (n=60)
Sampling Method: Non-Probability Sample
Enrollment: 195 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Study Retention | 6-12 months
  Proportion of participants completing the study
Daily survey/task adherence | 6-12 months
  Average completion of daily app-based surveys/tasks
Oura adherence | 6-12 months
  Average usage of the Oura smartring during study follow-up (minutes of daily device wear)
Empatica adherence | 6-12 months
  Average usage of the Empatica smartwatch during study follow-up (minutes of device on skin detection)
Bodyport adherence | 6-12 months
  Average usage of the Bodyport smartscale during study follow-up (number of weigh-ins)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Friend, MD, PhD, Principal Investigator — 4YouandMe
Locations (2):
- Mount Sinai, New York, New York, United States
- Nuffield Department of Population Health of Oxford University, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Subsets of the coded study data will be made accessible to researchers according to tiered permission:
  Internal Researchers (4YouandMe, Vector Institute, Evidation Health) will have access to all coded data.
  Collaboration Partners (Empatica, Bodyport, and Oura) will have access to a subset of coded data streams quarterly, with the exclusion of the video diary and any relative location data. Each partner will additionally have the data collected by their respective system.
  Clinical Collaborators will have access to the complete coded data set (with the exclusion of the video diary and any relative location data) at study end.
  De-identified data produced from this project will be shared broadly with qualified researchers through Sage Bionetworks Synapse. Only data from consenting participants will be shared through Sage Bionetworks Synapse and this will not include video diary data, relative location data or social media data.
Supporting Information: Study Protocol, ICF
Time Frame: Internal researchers will have access to all coded data during the full duration of the study. Consented participants' coded data will be available in the Synapse at Sage Bionetworks for selected researchers to access indefinitely, one year after study completion.
Access Criteria: Qualified Researcher
URL: https://www.synapse.org/